CLINICAL TRIAL: NCT01008631
Title: The Pharmacologic Profile of Sodium Thiosulfate in Renal Failure and Healthy
Brief Title: The Pharmacologic Profile of Sodium Thiosulfate in Renal Failure and Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Stefan Farese, Department of nephrology and hypertension, University of Berne, University of Berne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uehlinger-002
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Renal Failure
Keywords: renal failure; sodium Thiosulfate; pharmakokinetic
MeSH Terms: conditions — Renal Insufficiency | interventions — sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dialysis (Experimental): Two doses of sodium thiosulfate
  Interventions: Drug: Sodium thiosulfate
- healthy volunteer (Experimental): One dose of sodium thiosulfate
  Interventions: Drug: Sodium thiosulfate

INTERVENTIONS:
Drug: Sodium thiosulfate — 6g of Sodium Thiosulfate are applicated in a short infusion over a time of 5 min
  Other Names: Na2S2O3

SUMMARY:
The pharmacokinetics of sodium thiosulfate in humans with different degrees of renal failure and in healthy volunteers will be after two single shot applications.

DETAILED DESCRIPTION:
Two single shot applications of i.v. sodium thiosulfate will be given to dialysis patients. One application will be given immediately before a dialysis session and the second dose will be given after the consecutive dialysis session.

In healthy volunteers sodium thiosulfate will be given only once. In both groups, dialysis patients and healthy volunteers, blood and urinary/dialysate samples will be collected at defined time points.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer or patient with renal failure

Exclusion Criteria:

* pregnancy
* withdrawal of consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Elimination half life in dependence of the degree of renal failure | 0, 15, 30, 60, 180 minutes and 24 hours after application

SECONDARY OUTCOMES:
Changes in acid-base parameter after application of sodium thiosulfate | 0, 15, 30, 60, 180 minutes and 24 hours after application

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Farese, MD, Principal Investigator — University of Berne
Locations (1):
- Department of Nephrology and Hypertension, University of Berne, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Farese S, Stauffer E, Kalicki R, Hildebrandt T, Frey BM, Frey FJ, Uehlinger DE, Pasch A. Sodium thiosulfate pharmacokinetics in hemodialysis patients and healthy volunteers. Clin J Am Soc Nephrol. 2011 Jun;6(6):1447-55. doi: 10.2215/CJN.10241110. Epub 2011 May 12. PMID 21566113